CLINICAL TRIAL: NCT06680830
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of NEU-411 in Companion Diagnostic-Positive Participants With Early Parkinson's Disease
Brief Title: A Phase 2 Study of NEU-411 in Companion Diagnostic-Positive Participants With Early Parkinson's Disease
Acronym: NEULARK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neuron23 Inc. (Industry)
Collaborators: Qiagen Manchester Limited (Unknown); Roche Diagnostic Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEU-411-PD201
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease; Parkinson; Idiopathic Parkinson Disease; Early Parkinson Disease (Early PD); Parkinson Disease, Idiopathic
Keywords: Early PD; Parkinsons; Parkinsons Disease; Idiopathic Parkinsons Disease; leucine-rich repeat kinase 2; PD; NEULARK; LRRK2
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Sponsor is also masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (2):
- NEU-411 (Experimental): Orally-administered NEU-411
  Interventions: Drug: NEU-411
- Placebo (Placebo Comparator): Orally-administered matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NEU-411 — NEU-411, a potent, selective, orally bioavailable, highly permeable, brain penetrant, small molecule inhibitor of LRRK2 activity
  Arms: NEU-411
Other: Placebo — Orally-administered matched placebo
  Arms: Placebo

SUMMARY:
The goal of this Phase 2 clinical trial is to investigate the efficacy and safety of NEU-411 in men and women aged 40-80 years with early Parkinson's Disease (PD) who have predicted elevations in the activity of the "leucine-rich repeat kinase 2" ("LRRK2" for short) pathway based on their genetic profile. A DNA test will be used to identify the "LRRK2-driven" population with predicted elevation in the LRRK2 pathway.

Participants will:

• Take NEU-411 or placebo every day for 52 weeks

DETAILED DESCRIPTION:
NEU-411-PD201 is a Phase 2, randomized, placebo-controlled, proof-of-concept study in participants with early Parkinson's Disease (PD) who have LRRK2-driven PD as measured by an investigational companion diagnostic genetic test (CDx). The study will evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of NEU-411, an orally-administered, potent, selective, bioavailable, highly permeable, brain penetrant, small molecule inhibitor of LRRK2 activity as compared to placebo.

After participants are screened for inclusion in the study, approximately 150 participants will be randomized in a 1:1 allocation ratio to NEU-411 30 mg once per day or placebo for a 52-week treatment period. A safety follow-up visit will occur 2 weeks after the last treatment visit.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40-80 years at time of screening, inclusive
2. Diagnosis of clinically established or clinically probable Parkinson's Disease (PD)
3. LRRK2-driven PD using the investigational companion diagnostic genetic test (CDx)
4. Modified Hoehn and Yahr (mH&Y) of 1 to 2.5

Exclusion Criteria:

1. Secondary or atypical parkinsonian syndromes
2. Uncontrolled diabetes mellitus with hemoglobin A1c (HbA1c) >8%
3. Other significant medical conditions (as determined by medical history, examination, or clinical investigations at screening)

Additional inclusion and exclusion criteria are outlined in the full study protocol.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Roche digital biomarker score using the Roche Parkinson's Disease application (v3.0) compared to placebo | From enrollment to the end of treatment at 52 weeks
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) compared to placebo | From enrollment to the end of study at 54 weeks

SECONDARY OUTCOMES:
Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 52 weeks
  Change from baseline to Week 52 in motor function/nonmotor as measured by Movement Disorder Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS)

CONTACTS AND LOCATIONS:
Overall Officials: Fatta B Nahab, MD, FAAN FANA, Principal Investigator — Neuron23 Inc.
Locations (64):
- United States (43):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - Neuro-Pain Medical Center, Fresno, California
  - University of California, Irvine, Irvine, California
  - University of California, Los Angeles, Los Angeles, California
  - Esperanza Clinical, Murrieta, California
  - Parkinson's Research Centers of America - Palo Alto, Palo Alto, California
  - University of Colorado - Anschutz Medical Campus, Aurora, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - Neurology One, Orlando, Florida
  - USF Parkinson's & Movement Disorders Clinic, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Northwestern Medical Group, Department of Neurology, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Struthers Parkinson Center, Golden Valley, Minnesota
  - Cleveland Clinic, Las Vegas, Nevada
  - Northwell Health, Great Neck, New York
  - Icahn School of Medicine at Mount Sinai/Mount Sinai West, New York, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - The Ohio State University, Columbus, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Neurology Consultants of Dallas PA, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - University of Utah Movement Division, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - EvergreenHealth, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Italy (6):
  - IRCCS Ospedale San Raffaele (HSR) - Dipartimento Di Neurologia, Milan
  - Universita Degli Studi Della Campania "Luigi Vanvitelli" - Azienda Ospedaliera Universitaria, Napoli
  - Universita Degli Studi Di Padova - Azienda Ospedaliera Di Padova - Clinica Neurologica, Padua
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento Ospedaliero Di Santa Chiara, Pisa
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - San Raffaele Pisana, Rome
  - Fondazione Policilinico Universitario A Gemelli IRCCS, Rome
- Poland (4):
  - Centrum Medyczne Neuromed, Bydgoszcz
  - NZOZ Wielospecjalistyczna Poradnia Lekarska Synapsis Lech Szczechowski, Katowice
  - Pro Life Medica Sp. z o. o. ETA Lublin, Lublin
  - Insula Badania Sp. Z o.o., Warsaw
- Spain (7):
  - Policlinica Gipuzkoa - Centro de Investigacion Parkinson (CIP), San Sebastián, Donostia
  - Instituto de Investigacion Sanitaria Biocruces Bizkaia - Hospital Universitario Cruces, Barakaldo
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona (Hospital Clinic i Provincial) - Barnaclinic S.A., Barcelona
  - Universidad Autonoma de Madrid (UAM) - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario HM Puerta del Sur, Móstoles
  - Hospital Universitario Virgen del Rocio (HUVR) - Instituto de Biomedicina de Sevilla (IBIS), Seville
- United Kingdom (4):
  - St George's Hospital, University of London, London, England
  - University College London Hospitals NHS Foundation Trust, London, England
  - Clinical Aging Research Unit, Newcastle University, Newcastle upon Tyne, England
  - Ninewells Hospital and Medical School - NHS Tayside, Dundee, Scotland

IPD SHARING:
Plan to Share IPD: No